CLINICAL TRIAL: NCT07356687
Title: Effects of Dorsolateral Prefrontal Cortex rTMS Primed Dual-Task Gait Training on Walking and Cognitive Outcomes After Stroke: A Randomized Sham-Controlled Trial
Brief Title: Effects of rTMS Combined With Dual-Task Gait Training on Walking and Cognition After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Marco Yiu-Chung Pang, Chair professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20250731004
Record Dates: First submitted 2025-12-30; First posted 2026-01-21 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: Dual-task training; rTMS; Post-stroke rehabilitation; Cognitive-motor interference
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active rTMS with dual-task training (Experimental): Participants will receive rTMS targeting the DLPFC of the affected hemisphere immediately before each session of standardized dual-task gait training (12 sessions over 3 weeks)
  Interventions: Other: active rTMS with dual-task training
- sham rTMS with dual-task training (Active Comparator): Participants will receive sham rTMS (placebo stimulation) targeting the same DLPFC location immediately before each session of the same standardized dual-task gait training (12 sessions over 3 weeks).
  Interventions: Other: sham rTMS with dual-task training

INTERVENTIONS:
Other: active rTMS with dual-task training — Participants will receive active rTMS targeting the DLPFC of the affected hemisphere before each training session: 5 Hz, 90% resting motor threshold (RMT), 10-second trains with 30-second inter-train intervals, total 1,200 pulses (≈ 16 minutes) per session. Dual-task gait training will start within ~10 minutes after rTMS. The program includes 12 sessions over 3 weeks.
  Arms: active rTMS with dual-task training
Other: sham rTMS with dual-task training — Participants will receive sham rTMS delivered using the placebo side of the same coil at the same DLPFC target location and with identical session duration and procedures (≈ 16 minutes) before each training session. Dual-task gait training will start within ~10 minutes after sham stimulation. The program includes 12 sessions over 3 weeks.
  Arms: sham rTMS with dual-task training

SUMMARY:
This randomized, double-blind, placebo-controlled trial will investigate whether repetitive transcranial magnetic stimulation (rTMS) applied to the dorsolateral prefrontal cortex (DLPFC) can enhance the effects of dual-task gait training in people with chronic stroke. Participants will be randomly allocated to receive either active rTMS or sham rTMS immediately before the same standardized dual-task gait training program.

The intervention includes 12 sessions over 3 weeks. Outcomes will be assessed at baseline, immediately after training, and at 4-week follow-up. Co-primary outcomes are dual-task mobility and cognitive performance during walking, quantified using dual-task cost (DTC) for gait speed and cognitive-task performance during dual-task walking (e.g., Serial 7s; Shopping List Recall). Secondary outcomes include balance/mobility, community participation, mood/sleep measures, and fall incidence.

To explore mechanisms, prefrontal cortex activity during single- and dual-task walking will be recorded using functional near-infrared spectroscopy (fNIRS), and mediation analyses will examine whether changes in PFC activity explain intervention effects.

DETAILED DESCRIPTION:
Cognitive-motor interference after stroke can reduce walking safety and functional independence, especially during everyday dual-task situations. Dual-task gait training can improve performance, but response varies, potentially due to limitations in executive control and prefrontal network engagement. The DLPFC is central to attention and executive function; therefore, rTMS targeting the DLPFC may prime relevant neural circuits and improve responsiveness to subsequent dual-task training.

This study is a parallel-group, randomized, double-blind, placebo-controlled trial. Community dwelling adults with chronic unilateral stroke will be recruited and randomized 1:1. Participants and outcome assessors will be blinded.

Both groups will complete 12 supervised sessions over 3 weeks. In each session, participants will first receive either: Active rTMS to the DLPFC of the affected hemisphere (5 Hz; 90% resting motor threshold; total 1,200 pulses), or Sham rTMS using the placebo side of the coil with similar auditory sensations.

Dual-task gait training will begin shortly after stimulation. Training will combine functional walking/balance tasks with progressively challenging cognitive tasks (e.g., mental arithmetic, verbal fluency, working memory tasks, and a shopping-list recall task), with difficulty adjusted to participant ability.

Assessments will be conducted at baseline, post-intervention, and 4-week follow-up. Co-primary outcomes are DTC of gait speed and cognitive performance during dual-task walking.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ischemic or hemorrhagic hemispheric stroke
* Age ≥ 50 years

  -≥ 6 months post-stroke
* Medically stable
* Able to walk independently ≥ 1 minute (assistive device allowed)
* Able to follow commands
* mRS 1-3
* MoCA ≥ 22

Exclusion Criteria:

* Other neurological disorders
* Cerebellar/brainstem injury
* TMS contraindications (e.g., pacemaker, intracranial metal, seizure history, pregnancy)
* Contraindications to exercise (e.g., unstable angina)
* Severe aphasia (NIHSS item 9 ≥ 2)
* Pain/illness limiting performance
* Concurrent formal rehabilitation elsewhere
* RMT cannot be determined
* Fails TMS safety screening

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2026-01-21 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Dual-task cost (DTC) of walking speed (%) | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  Walking speed (m/s) measured during single-task walking and dual-task walking (walking + Serial 7s; walking + Shopping List Recall). DTC computed as (single-task - dual-task) / single-task × 100%; higher DTC indicates greater cognitive-motor interference. Speed will be averaged across three 45-s trials per condition.
Dual-task cost (DTC) of cognitive performance (%) | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  Cognitive performance recorded as number of correct responses during dual-task walking conditions:
  Serial 7s: number of correct subtractions during the 45-s trial Shopping List Recall: number of items correctly recalled immediately after the 45-s sitting/walking trial.
  DTC computed as (single-task - dual-task) / single-task × 100%; higher DTC indicates worse cognitive-motor interference. Values averaged across three trials per condition.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) time (seconds) | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  Time in seconds to complete: (1) standard TUG, and (2) cognitive dual-task TUG with serial 3 subtraction. Lower time indicates better functional mobility.
Mini-BESTest total score | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  Mini-BESTest total score assessing dynamic balance; higher score indicates better balance control.
Activities-specific Balance Confidence Scale (ABC) score | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  Self-reported balance confidence (0-100%); higher score indicates greater confidence during daily activities.
Fall incidence (number of falls) | During 6 months post-intervention follow-up
  Number of falls recorded using a fall diary and confirmed during scheduled follow-up contacts.
Stride length (cm) | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  Mean stride length during walking assessed using wearable sensors.
Reintegration to Normal Living Index (RNLI) score | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  RNLI score reflecting community participation and reintegration; higher score indicates better reintegration to normal living.
Cadence (steps/min) | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  Description: Mean cadence during gait, derived from wearable sensor data.
Double support time (%) | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  Percentage of gait cycle spent in double support.
Gait Speed (m/s) | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  The rate at which an individual covers distance while walking, typically measured in meters per second.
Foot Strike Angle (degrees) | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  The angle of the foot relative to the ground at the moment of initial contact.
Turns - Duration (seconds) | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  The time taken to complete a turn while walking.
Session-level perceived fatigue (0-10 rating) | Before and after each training session (3 weeks)
  Self-reported fatigue level rated on a 0-10 numerical scale, assessed immediately before and after each training session. Higher scores indicate greater perceived fatigue.
Number of participants with adverse events | During the 3-week intervention period
  Number of participants experiencing adverse events related to tms and dual-task gait training.

OTHER OUTCOMES:
Prefrontal cortex hemodynamic response (fNIRS HbO) during walking | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  Changes in bilateral prefrontal cortex oxyhemoglobin (HbO) measured by fNIRS during single- and dual-task walking; used as a mechanistic/mediator outcome.
Depression Anxiety Stress Scales-21 (DASS-21) subscale scores | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  Depression, Anxiety, and Stress subscale scores from DASS-21; higher scores indicate greater emotional distress.
Pittsburgh Sleep Quality Index (PSQI) global score | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  PSQI global score assessing sleep quality; higher score indicates poorer sleep quality.
Fugl-Meyer Assessment-Lower Extremity (FMA-LE) score | Baseline (pre-intervention), 1-week post-intervention (Week 4), and 4-week post-intervention follow-up (Week 8)
  FMA-LE motor score (0-34); higher score indicates better lower-limb motor recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, HongKong, Hong Kong

IPD SHARING:
Plan to Share IPD: No